CLINICAL TRIAL: NCT00834522
Title: A Single-Dose, Comparative Bioavailability Study of Two Formulations of Granisetron 1 mg Tablets Under Fed Conditions
Brief Title: Granisetron 1 mg Tablets, Non-fasting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2005-1021
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Granisetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Granisetron (Experimental): Granisetron 2 x 1 mg Tablet (test) dosed in first period followed by Kytril® 2 x 1 mg Tablet (reference) dosed in second period
  Interventions: Drug: Granisetron hydrochloride 1 mg tablets
- Kytril® (Active Comparator): Kytril® 2 x 1 mg Tablet (reference) dosed in first period followed by Granisetron 2 x 1 mg Tablet (test) dosed in second period
  Interventions: Drug: Kytril® 1 mg tablets

INTERVENTIONS:
Drug: Granisetron hydrochloride 1 mg tablets — 2 x 1 mg, single dose non-fasting
  Arms: Granisetron
Drug: Kytril® 1 mg tablets — 2 x 1 mg, single dose non-fasting
  Arms: Kytril®

SUMMARY:
The objective of this study is to evaluate the comparative bioavailability between granisetron hydrochloride 1 mg tablets (Teva Pharmaceuticals USA) and Kytril® 1 mg tablets (Roche, USA), after a single-dose in health subjects under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking, male and female subjects, 18 years of age or older.
* BMI ≥ 19 and ≤ 30.
* No significant diseases or clinically significant findings in a physical - examination.
* No clinically significant abnormal laboratory values.
* No clinically significant findings in the 12-lead electrocardiogram (ECG).
* No clinically significant findings from the vital signs measurement.
* Be informed of the nature of the study and given written consent prior to receiving any study procedure.

Negative for:

* HIV.
* Hepatitis B surface antigen and Hepatitis C antibody.
* Urine drugs of abuse test (marijuana, amphetamines, barbiturates, cocaine, opiates, benzodiazepines and methadone).
* Urine cotinine test.
* Serum HCG consistent with pregnancy (females only).

Females who participate in this study are:

* unable to have children (e.g. post-menopausal, tubal ligation, hysterectomy) OR
* willing to remain abstinent [not engage in sexual intercourse] OR
* willing to use an effective method of double-barrier birth control [partner using condom and female using diaphragm, contraceptive sponge, spermicide or IUD]
* Females who participate in this study are not pregnant and/or non-lactating.

Exclusion Criteria:

* Known history or presence of any clinically significant medical condition.
* Known or suspected carcinoma.
* On a special diet within 4 weeks prior to drug administration (e.g. liquid, protein, raw food diet).
* Participated in another clinical trial or received an investigational product within 30 days prior to drug administration.
* Donated up to 250 mL of blood within the previous 30 days OR Donated from 251 to 500 mL of blood in the previous 45 days OR Donated more than 500 mL of blood in the previous 56 days (based on the Canadian Blood Services guideline for blood donation).
* Females taking oral or transdermal hormonal contraceptives within 14 days preceding period 1 dosing OR females having taken implanted or injected hormonal contraceptives within 6 months prior to period 1 dosing.
* Requirement of any non-topical medication (prescription and/or over-the-counter) on a routine basis.
* Difficulty fasting or consuming the standard meals.
* Do not tolerate venipuncture.
* Unable to read or sign the ICF.

Known history or presence of:

* Hypersensitivity or idiosyncratic reaction to granisetron hydrochloride and/or any other drug substances with similar activity.
* Alcoholism within the last 12 months.
* Drug dependence and/or substance abuse.
* Use of tobacco or nicotine-containing products, within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-07; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xueyu (Eric) Chen, M.D., Ph. D., Principal Investigator — Pharma Medica
Locations (1):
- Pharma Medica Research Inc, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Granisetron (Test) First: Granisetron 2 x 1 mg Tablet (test) dosed in first period followed by Kytril® 2 x 1 mg Tablet (reference) dosed in second period
- Kytril® (Reference) First: Kytril® 2 x 1 mg Tablet (reference) dosed in first period followed by Granisetron 2 x 1 mg Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Granisetron (Test) First | Kytril® (Reference) First
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0
Period: Washout
Arm/Group | Granisetron (Test) First | Kytril® (Reference) First
Started | 40 | 40
Completed | 37 | 39
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Period: Second Intervention
Arm/Group | Granisetron (Test) First | Kytril® (Reference) First
Started | 37 | 39
Completed | 37 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Granisetron (Test) First | Kytril® (Reference) First | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 22 | 25 | 47
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 34 | 28 | 62
  Black | 6 | 10 | 16
  Asian | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration)
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Granisetron: Granisetron 2 x 1 mg Tablet (test) dosed in either period
- Kytril®: Kytril® 2 x 1 mg Tablet (reference) dosed in either period
Arm/Group | Granisetron | Kytril®
Number analyzed (Participants) | 76 | 76
ng/mL | 10.4016 (3.4598) | 10.1061 (3.2848)
Statistical Analysis 1: Comparison: Granisetron vs Kytril®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Geometric Test/Ref Ratio x 100 = 103.79, 90% CI [99.40 to 108.37] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf [Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)]
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Granisetron | Kytril®
Number analyzed (Participants) | 76 | 76
ng*h/mL | 130.3581 (68.2310) | 126.9140 (72.9558)
Statistical Analysis 1: Comparison: Granisetron vs Kytril®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Geometric Test/Ref Ratio x 100 = 104.37, 90% CI [97.04 to 112.25] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t [Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)]
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Granisetron | Kytril®
Number analyzed (Participants) | 76 | 76
ng*h/mL | 127.6581 (66.0753) | 124.4104 (70.2712)
Statistical Analysis 1: Comparison: Granisetron vs Kytril®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Geometric Test/Ref Ratio x 100 = 104.22, 90% CI [96.90 to 112.08] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.